CLINICAL TRIAL: NCT07399366
Title: Effect of a Film-Based "Medical Education and Social Justice" Elective on Medical Students' Alexithymia Levels and Empathy Skills: A Nonrandomized Controlled Pretest-Posttest Study
Brief Title: Film-Based Medical Education and Social Justice Course: Effects on Alexithymia and Empathy in Medical Students
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Çanakkale Onsekiz Mart University (Other)
Responsible Party: Principal Investigator, Mustafa Onur Yurdal, PhD, Curriculum Specialist, Çanakkale Onsekiz Mart University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2025-YÖNP-0418
Record Dates: First submitted 2026-02-03; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Alexithymia; Empathy Skills; Education, Medical; Social Justice Advocacy; Health Equity
Keywords: Film-based education; Cinema in medical education; CineMedicine; Narrative medicine; Social justice education
MeSH Terms: conditions — Affective Symptoms; Narrative Medicine

STUDY DESIGN:
Intervention Model Description: Nonrandomized allocation due to elective self-selection (students enroll in the course by choice); contemporaneous comparison group not enrolled.
Who Masked: Outcomes Assessor
Masking Description: Outcomes Assessor: Scenario-based empathy responses are scored by independent raters who are blinded to group assignment (elective vs control) and time point (T0 vs T1). Responses are de-identified and labeled with coded participant IDs prior to scoring. Unblinding occurs only after scoring is completed.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Film-Based Medical Education and Social Justice Elective (Experimental): Participants enrolled in the elective "Film-Based Medical Education and Social Justice" course. The course is delivered over one semester (~14 weeks) and uses selected films/film clips with structured group discussion and reflection activities.
  Interventions: Behavioral: Film-Based Medical Education and Social Justice Elective
- No Course / Usual Curriculum (No Intervention): Participants who do not enroll in the elective course during the same period and continue usual curriculum without additional sessions.

INTERVENTIONS:
Behavioral: Film-Based Medical Education and Social Justice Elective — A 14-week elective course (approximately 2 hours/week) using selected films/film clips with structured group discussion and reflective activities/journaling.
  Other Names: Film-Based Medical Education and Social Justice Course
  Arms: Film-Based Medical Education and Social Justice Elective

SUMMARY:
This study will examine whether a 14-week elective course that uses films and guided discussion on social justice in health care can improve medical students' empathy skills and reduce alexithymia (difficulty recognizing and describing emotions). Approximately 50 volunteer medical students will participate. Students who choose the elective course will form the intervention group, and students who do not take the course will form a comparison group. All participants will complete the same questionnaires/assessments at the beginning and at the end of the semester. The main goal is to compare changes in empathy and alexithymia scores between the two groups.

DETAILED DESCRIPTION:
This is a prospective, nonrandomized controlled pretest-posttest study conducted at Canakkale Onsekiz Mart University Faculty of Medicine. Participants are volunteer medical students (≥18 years). The intervention group consists of students who enroll in the elective course, and the comparison group consists of students from the same student population who do not enroll during the same period.

Data will be collected at two time points: baseline prior to the start of the elective period (T0) and immediately after the end of the elective period (T1, approximately 14 weeks later). At each time point, participants will complete the study instruments administered in a standardized manner. In the intervention group, reflective journals will also be collected throughout the course period to support qualitative interpretation of findings.

The primary analysis will compare within-group change from T0 to T1 and between-group differences in change scores. Descriptive statistics will summarize participant characteristics. Depending on data distribution, paired tests and independent-group tests (or their nonparametric equivalents) will be used for continuous outcomes. Multivariable models may be used to adjust for baseline differences (e.g., class year) if imbalance is observed. Missing data will be handled using a predefined approach (e.g., complete-case analysis with sensitivity checks). No clinical procedures or medical treatments are involved.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled medical student at Canakkale Onsekiz Mart University Faculty of Medicine, registered in Year 1, 2, or 3 during the study period.
* Age 18 years or older.
* Provides written/electronic informed consent after being informed about the study.
* For the intervention arm: enrolled in the elective "Film-Based Medical Education and Social Justice" course.
* For the control arm: from the same academic year/cohort during the same period and not enrolled in the elective course.
* Willing and able to complete both baseline (T0) and end-of-course (T1) assessments (has sufficient cognitive/communication ability to complete questionnaires).

Exclusion Criteria:

* Does not provide consent or withdraws consent at any stage.
* Younger than 18 years.
* Does not complete at least one of the two assessments (T0 or T1).
* Leaves critical sections of the questionnaires/assessments largely blank (e.g., substantial missing items on TAS-20 or incomplete scenario responses preventing scoring).
* Duplicate/duplicate submission (more than one form from the same participant for the same assessment).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-02-16 (Estimated); Primary Completion 2026-06-20 (Estimated); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
Toronto Alexithymia Scale (TAS-20) Total and Subscale Scores (Change) | Baseline (T0) and end of course (T1, approximately 14 weeks)
  Change in TAS-20 total score and subscale scores (Difficulty Identifying Feelings, Difficulty Describing Feelings, Externally Oriented Thinking). Higher scores indicate higher alexithymia.
Scenario-Based Empathy Skills Total Score and Rubric Subscores (Change) | Baseline (T0) and end of course (T1, approximately 14 weeks)
  Change in total empathy skills score derived from responses to study-developed scenarios scored with a rubric based on Dökmen's staged empathy classification; includes rubric subscores/levels if applicable.

SECONDARY OUTCOMES:
Association Between Change in TAS-20 and Change in Empathy Score | From baseline (T0) to end of course (T1, approximately 14 weeks)
  Correlation/association between ΔTAS-20 (T1-T0) and ΔEmpathy (T1-T0) (Pearson or Spearman depending on distribution).

OTHER OUTCOMES:
Reflective Journal Themes (Intervention Group Only) | After each session during the course period (approximately 14 weeks); analyzed after T1
  De-identified reflective journals collected after sessions will be analyzed using thematic/content analysis to contextualize and deepen interpretation of quantitative findings.

CONTACTS AND LOCATIONS:
Overall Officials: Mustafa Onur Yurdal, PhD, Study Chair — Çanakkale Onsekiz Mart University
Locations (1):
- Faculty of Medicine, Çanakkale, Çanakkale, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
De-identified individual participant data (IPD) underlying the results reported in publications (e.g., TAS-20 total/subscale scores and scenario-based empathy scores at T0 and T1) will be made available to qualified researchers upon reasonable request. Data will be shared after publication of the primary results, for up to 5 years. Requests will be reviewed by the study team and may require a data use agreement. Shared datasets will be de-identified and will not include direct identifiers; access will be limited to the minimum necessary to protect participant confidentiality.

REFERENCES:
- [Result] Bagby RM, Parker JD, Taylor GJ. The twenty-item Toronto Alexithymia Scale- I. J Psychosom Res. 1994;38(1):23-32. PMID: 8126686. doi: 10.1016/0022-3999(94)90005-1. Law M, Kwong W, Friesen F, Veinot P, Ng SL. The current landscape of television and movies in medical education. Perspect Med Educ. 2015;4(5):218-224. doi: 10.1007/s40037-015-0205-9. Lumlertgul N, Kijpaisalratana N, Pityaratstian N, Wangsaturaka D. Cinemeducation: A pilot student project using movies to help students learn medical professionalism. Med Teach. 2009;31(7):e327-e332. PMID: 19811142. doi: 10.1080/01421590802637941. Rueb M, Siebeck M, Rehfuess EA, Pfadenhauer LM. Cinemeducation in medicine: a mixed methods study on students' motivations and benefits. BMC Med Educ. 2022;22:172. doi: 10.1186/s12909-022-03240-x. Salajegheh M, Sohrabpour AA, Mohammadi E. Exploring medical students' perceptions of empathy after cinemeducation based on Lev Vygotsky's theory. BMC Med Educ. 2024;24:94. doi: 10.1186/s12909-024-05084-z.
- See also: Course Syllabus — https://ubys.comu.edu.tr/AIS/OutcomeBasedLearning/Home/CourseDetail?=undefined&isElectiveCourse=true&isIntegratedCourse=false&courseId=!xBBx!H44nwS!xBBx!!xBBx!4ZZM92m!xDDx!xlnjw!xGGx!!xGGx!&curriculumId=t8XuNQUexfCE4FCNR!xBBx!suHg!xGGx!!xGGx!&apid=Lm3u4Yh8tC2r3etb20o5EA!xGGx!!xGGx!&eqd=10602&progName=Rekt%C3%B6rl%C3%BCk%20-%20T%C4%B1p%20Fak%C3%BCltesi%20/%20T%C4%B1p--Lisans%20-%20Normal%20%C3%96%C4%9Fretim&culture=en-US&year=2023